CLINICAL TRIAL: NCT02983604
Title: A Phase 1b/2 Study of GS-5829 in Combination With Fulvestrant or Exemestane in Subjects With Advanced Estrogen Receptor Positive, HER2 Negative-Breast Cancer
Brief Title: GS-5829 in Combination With Fulvestrant or Exemestane in Women With Advanced Estrogen Receptor Positive, HER2 Negative-Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-350-1937; 2016-002365-63 (EudraCT Number)
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Advanced Estrogen Receptor Positive HER2- Breast Cancer
Keywords: Exemestane; Aromasin; Fulvestrant; Faslodex; Breast Cancer; HER 2-; Estrogen receptor positive
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GS-5829 + exemestane (Phase 1b) (Experimental): Participants will be sequentially enrolled at progressively higher dose levels of GS-5829 (up to 9 mg) in combination with exemestane and may continue with treatment until disease progression, unacceptable toxicity, withdrawal of consent, or death, whichever comes first.
  Interventions: Drug: GS-5829; Drug: Exemestane
- GS-5829 + fulvestrant (Phase 1b) (Experimental): Participants will be sequentially enrolled at progressively higher dose levels of GS-5829 (up to 9 mg) in combination with fulvestrant and may continue with treatment until disease progression, unacceptable toxicity, withdrawal of consent, or death, whichever comes first.
  Interventions: Drug: GS-5829; Drug: Fulvestrant
- GS-5829 + fulvestrant (Phase 2) (Experimental): Participants will receive GS-5829 (dose determined from Phase 1b) + fulvestrant until disease progression, unacceptable toxicity, withdrawal of consent, or death, whichever comes first.
  Interventions: Drug: GS-5829; Drug: Fulvestrant
- Fulvestrant (Phase 2) (Active Comparator): Participants will receive fulvestrant alone until disease progression, unacceptable toxicity, withdrawal of consent, or death, whichever comes first.
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: GS-5829 — Tablet(s) administered orally once daily
  Arms: GS-5829 + exemestane (Phase 1b); GS-5829 + fulvestrant (Phase 1b); GS-5829 + fulvestrant (Phase 2)
Drug: Exemestane — 25 mg tablet administered orally once daily (or in accordance with locally approved labeling)
  Other Names: Aromasin®
  Arms: GS-5829 + exemestane (Phase 1b)
Drug: Fulvestrant — Administered every 28 days (± 3 days) intramuscularly in accordance with locally approved labeling
  Participants initiating fulvestrant on Cycle 1 Day 1 and have not received any prior dose of fulvestrant will receive a single additional dose of fulvestrant on Cycle 1 Day 15.
  Other Names: Faslodex®
  Arms: Fulvestrant (Phase 2); GS-5829 + fulvestrant (Phase 1b); GS-5829 + fulvestrant (Phase 2)

SUMMARY:
The primary objectives of the Phase 1b Dose Escalation part of this study are to characterize the safety and tolerability of GS-5829 in combination with exemestane or fulvestrant and to determine the maximum tolerated dose (MTD) or the recommended Phase 2 dose of GS-5829 in combination with fulvestrant in women with advanced estrogen receptor positive, HER2-negative (ER+/HER2-) breast cancer.

The primary objective of the Randomized Phase 2 Dose Expansion portion of this study is to evaluate the efficacy of GS-5829 in combination with fulvestrant compared to fulvestrant alone in women with advanced ER+/HER2- breast cancer.

This study was terminated early and the Phase 2 portion of the study was not conducted.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer with evidence of metastatic or locally advanced disease not amenable to resection or radiation therapy with curative intent and who have progressed during treatment with at least one prior hormonal therapy

  * Phase 1b Dose Escalation - Individuals may have had unlimited prior hormonal therapy and a total of 2 prior chemotherapy regimens (adjuvant chemotherapy is considered 1 regimen). Individuals may have progressed on fulvestrant or exemestane.
  * Randomized Phase 2 Dose Expansion - Individuals may have disease progression during treatment or within 12 months of completion of endocrine therapy (tamoxifen, and/or AI) in the adjuvant setting, or disease progression during treatment with endocrine therapy (tamoxifen, AI or CDK4/6 inhibitor plus AI) for advanced/metastatic disease. Individuals may have had unlimited prior hormonal therapy, but must be naive to fulvestrant in the metastatic setting. A total of 2 prior chemotherapies are allowed, however, only one for metastatic disease is permitted.
* Documentation of ER positive (≥ 1% positive stained cells by local standards) based on the most recent tumor biopsy, unless bone-only disease
* Documented HER2-negative tumor based on local testing on most recent tumor biopsy (immunohistochemistry score 0/1+ or negative by in situ hybridization HER2/CP17 ratio < 2 or for single probe assessment HER2 copy number < 4)
* Post-, pre- or peri-menopausal women considered to be in the post-menopausal state as defined by one of the following:

  * Age ≥ 60 years
  * Age < 60 years and cessation of regular menses for at least 12 consecutive months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression and serum estradiol and follicle-stimulating hormone (FSH) level within the post-menopausal range
  * Prior bilateral oophorectomy
  * Pre-/peri-menopausal women can be enrolled if amenable to be treated with the luteinizing-hormone releasing hormone (LHRH) agonist, goserelin. Individuals must have commenced treatment with goserelin or an alternative LHRH agonist at least 4 weeks prior to Cycle 1 Day 1 (C1D1). If individuals have received an alternative LHRH agonist prior to study entry, they must switch to goserelin on or before Cycle 1 Day 1 (C1D1) for the duration of the study
* Measurable disease defined per RECIST v. 1.1, or bone-only disease must have a lytic or mixed lytic blastic lesion that can be accurately assessed by computed tomography (CT) or magnetic resonance imaging (MRI). Individuals with bone-only disease and blastic-only metastases are not eligible
* All acute toxic effects of any prior antitumor therapy resolved to Grade ≤ 1 before the start of study drug dosing (with the exception of alopecia [Grade 1 or 2 permitted] and neurotoxicity [Grade 1 or 2 permitted])
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1
* Life expectancy of ≥ 3 months, in the opinion of the investigator
* Adequate organ function defined as follows:

  * Hematologic: Platelets ≥ 100 x 10^9/L; Hemoglobin ≥ 9.0 g/dL; absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (without platelet transfusion or any granulocytic growth factors within previous 7 days of the hematologic laboratory values obtained at screening visit)
  * Hepatic: aspartate transaminase (AST) / alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN) (if liver metastases are present, ≤ 5 x ULN); total or conjugated bilirubin ≤ 1.5 x ULN
  * Renal: Serum Creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 60 mL/min as calculated by the Cockroft-Gault method
* Coagulation: International Normalized Ratio (INR) ≤ 1.2
* Negative serum pregnancy test
* Females of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception as described in the study protocol
* Females who are nursing must agree to discontinue nursing before the first dose of GS-5829
* Able and willing to provide written informed consent to participate in the study

Key Exclusion Criteria:

* History or evidence of clinically significant disorder, condition, or disease that, in the opinion of the investigator or the Gilead medical monitor would pose a risk to individual safety or interfere with the study evaluations, procedures, or completion
* Known brain metastasis or leptomeningeal disease (Note: if treated and stable at least 6 months prior to enrollment, individual is eligible).
* Uncontrolled intercurrent illness including, but not limited to, active uncontrolled infection, active or chronic bleeding event within 28 days prior to C1D1, uncontrolled cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements as judged by treating physician
* Myocardial infarction, symptomatic congestive heart failure (New York Heart Association Classification > Class II), unstable angina, or serious uncontrolled cardiac arrhythmia within the last 6 months of C1D1
* Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (i.e., larger than what is required for placement of central venous access, percutaneous feeding tube) within 28 days of C1D1
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of GS-5829, including any unresolved nausea, vomiting, or diarrhea that is Common Terminology Criteria for Adverse Events (CTCAE) Grade > 1
* Minor surgical procedure(s) within 7 days of enrollment or randomization, or not yet recovered from prior surgery (placement of central venous access device, fine needle aspiration, or endoscopic biliary stent ≥ 1 day before enrollment or randomization is acceptable)
* History of a concurrent or second malignancy, except for: adequately treated local basal cell or squamous cell carcinoma of the skin; cervical carcinoma in situ; superficial bladder cancer; adequately treated Stage 1 or 2 cancer currently in complete remission; any other cancer that has been in complete remission for ≥ 5 years
* Anti-tumor therapy (chemotherapy, chemoradiation, radiation, antibody therapy, molecular targeted therapy) within 21 days or 5 half-lives whichever is longer, of C1D1 (6 weeks for nitrosoureas, mitomycin C, or molecular agents with t1/2 > 10 days); 5 half-lives of any investigational drug; concurrent use of goserelin for pre-/peri-menopausal breast cancer and exemestane or fulvestrant per the protocol are permitted
* History of long QT syndrome or whose corrected QT interval (QTc) measured (Fridericia method) at screening is prolonged (> 470 ms). Individuals who screen fail due to this criterion are not eligible to be re-screened
* Prior exposure to any bromodomain (BET) inhibitors
* Known hypersensitivity to the study drugs (GS 5829, fulvestrant or exemestane), the metabolites, or formulation excipients
* Immunotherapy within 6 months of C1D1
* Evidence of bleeding diathesis or clinically significant bleeding, within 28 days of C1D1 or history of hemoptysis of > 2.5 mL/1 teaspoon within 6 months of C1D1
* Anticoagulation/antiplatelet therapy within 7 days of C1D1, including acetylsalicylic acid, low molecular weight heparin, or warfarin
* Known human immunodeficiency virus (HIV) infection
* Hepatitis B surface Antigen (HBsAg) positive
* Hepatitis C virus (HCV) antibody positive with HCV RNA positive
* Use of moderate/strong cytochrome P450 (CYP)3A4 inhibitors or moderate/strong CYP3A4 inducers within 2 weeks prior to C1D1
* History of high grade esophageal or gastric varices

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- United States (6):
  - Stanford Women's Cancer Center, Stanford, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Allina Health, Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor University Medical Center, Houston, Texas
  - Medical Oncology Associates, PS (dba Summit Cancer Centers), Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 10 January 2017. The last study visit occurred on 19 July 2018.
Pre-assignment Details: 17 participants were screened.
Groups:
- GS-5829 4 mg + Exemestane: GS-5829 4 mg tablets once daily + exemestane 25 mg tablet once daily
- GS-5829 4 mg + Fulvestrant: GS-5829 4 mg tablets once daily + fulvestrant 500 mg administered intramuscularly every 28 days (± 3 days)
- GS-5829 6 mg + Fulvestrant: GS-5829 6 mg tablets once daily + fulvestrant 500 mg administered intramuscularly every 28 days (± 3 days)
- GS-5829 9 mg + Fulvestrant: GS-5829 9 mg tablets once daily + fulvestrant 500 mg administered intramuscularly every 28 days (± 3 days)
Period: Overall Study
Arm/Group | GS-5829 4 mg + Exemestane | GS-5829 4 mg + Fulvestrant | GS-5829 6 mg + Fulvestrant | GS-5829 9 mg + Fulvestrant
Started | 4 | 3 | 4 | 3
Completed | 4 | 3 | 3 | 3
Not Completed | 0 | 0 | 1 | 0
Not completed — Enrolled but not Treated | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who were enrolled and received at least 1 dose of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | GS-5829 4 mg + Exemestane | GS-5829 4 mg + Fulvestrant | GS-5829 6 mg + Fulvestrant | GS-5829 9 mg + Fulvestrant | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (4.50) | 61.3 (7.51) | 63.0 (9.54) | 65.0 (12.29) | 61.9 (7.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 3 | 13
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 3 | 3 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 3 | 3 | 12
  Other | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b Dose Escalation: Number of Participants Experiencing Dose Limiting Toxicities (DLTs) Through Day 28 at Each Dose Level of GS-5829
Description: A DLT was a toxicity as defined below:
  * Grade ≥ 4 neutropenia
  * Grade ≥ 3 neutropenia with fever
  * Grade ≥ 3 thrombocytopenia
  * Grade ≥ 2 bleeding (e.g., gastrointestinal, respiratory, epistaxis, purpura)
  * Grade ≥ 3 or higher non-hematologic toxicity, except:
    * Grade 3 nausea or emesis with maximum duration of 48 hours on adequate medical therapy
    * Grade 3 diarrhea which persists for < 72 hours in the absence of adequate medical therapy
  * Grade ≥ 2 non-hematologic treatment-emergent adverse event (TEAE) that in the opinion of the investigator is of potential clinical significance such that further dose escalation would expose participants to unacceptable risk
  * Treatment interruption of ≥ 7 days due to unresolved toxicity
  * Grade 3 or Grade 4 elevation in aspartate transaminase (AST) or alanine transaminase (ALT) associated with a Grade 2 elevation in bilirubin that is at least possibly related to study drug
Time Frame: Baseline up to 28 days
Population: The DLT Analysis Set included all participants in the Safety Analysis Set who completed all treatment and safety procedures through Day 28, inclusive, or experienced a DLT prior to Day 28, exclusive.
Measure: Count of Participants; unit: Participants
Groups:
- GS-5829 4 mg + Fulvestrant: GS-5829 4 mg tablets once daily + fulvestrant 500 mg administered intramuscularly on Days 1, 15, and 29, and then every 28 days (or in accordance with locally approved labeling)
- GS-5829 6 mg + Fulvestrant: GS-5829 6 mg tablets once daily + fulvestrant 500 mg administered intramuscularly on Days 1, 15, and 29, and then every 28 days (or in accordance with locally approved labeling)
- GS-5829 9 mg + Fulvestrant: GS-5829 9 mg tablets once daily + fulvestrant 500 mg administered intramuscularly on Days 1, 15, and 29, and then every 28 days (or in accordance with locally approved labeling)
Arm/Group | GS-5829 4 mg + Exemestane | GS-5829 4 mg + Fulvestrant | GS-5829 6 mg + Fulvestrant | GS-5829 9 mg + Fulvestrant
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants | 1 | 0 | 0 | 0

2. Primary Outcome: Randomized Phase 2 Dose Expansion: Progression-Free Survival
Description: Progression-Free Survival (PFS) was defined as the interval from date of randomization to the earlier of the first documented confirmed disease progression or death from any cause.
Time Frame: Baseline up to 2 years
Population: As the study was terminated prior to the Phase 2 portion of the study, no participants were enrolled in the Phase 2 portion of the study and data was not collected for this endpoint.
Arm/Group | GS-5829 4 mg + Exemestane | GS-5829 4 mg + Fulvestrant | GS-5829 6 mg + Fulvestrant | GS-5829 9 mg + Fulvestrant
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Phase 1b Dose Escalation: Pharmacokinetic (PK) Parameter: Cmax of GS-5829
Description: Cmax is defined as the maximum observed concentration of drug.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours postdose on Days 1 and 15
Population: The PK Analysis Set included all enrolled participants who received at least 1 dose of study drug and have at least 1 nonmissing postdose concentration value reported by the PK laboratory, excluding participants who received concomitant medications prohibited in this study. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GS-5829 4 mg + Exemestane | GS-5829 4 mg + Fulvestrant | GS-5829 6 mg + Fulvestrant | GS-5829 9 mg + Fulvestrant
Number analyzed (Participants) | 4 | 3 | 3 | 2
ng/mL
  Day 1 | 318.25 (107.844) | 247.00 (3.464) | 244.00 (9.000) | 518.00 (60.811)
  Day 15: number analyzed (Participants) | 3 | 3 | 3 | 2
  Day 15 | 389.666 (105.6424) | 370.333 (52.5483) | 375.666 (67.0919) | 634.000 (46.6690)

4. Secondary Outcome: Phase 1b Dose Escalation: PK Parameter: AUCtau of GS-5829
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours postdose on Day 15
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | GS-5829 4 mg + Exemestane | GS-5829 4 mg + Fulvestrant | GS-5829 6 mg + Fulvestrant | GS-5829 9 mg + Fulvestrant
Number analyzed (Participants) | 3 | 3 | 3 | 2
h*ng/mL | 4989.809 (1655.8737) | 5218.820 (1326.2407) | 3937.709 (667.4396) | 7638.847 (938.3444)

5. Secondary Outcome: Randomized Phase 2 Dose Expansion: Overall Safety Profile as Assessed by the Percentage of Participants Experiencing Any Adverse Events (AEs), Grade 3 or 4 AEs, Treatment-Related AEs, or Abnormalities in Laboratory Tests or Electrocardiograms
Time Frame: Baseline up to 2 years
Population: as for outcome 2
Arm/Group | GS-5829 4 mg + Exemestane | GS-5829 4 mg + Fulvestrant | GS-5829 6 mg + Fulvestrant | GS-5829 9 mg + Fulvestrant
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Randomized Phase 2 Dose Expansion: Overall Response Rate
Description: Overall response rate (ORR) was defined as the proportion of participants who achieve complete response (CR) or partial response (PR), based on Response Evaluation Criteria in Solid Tumors (RECIST) v. 1.1 study progression criteria.
Time Frame: Baseline up to 2 years
Population: as for outcome 2
Arm/Group | GS-5829 4 mg + Exemestane | GS-5829 4 mg + Fulvestrant | GS-5829 6 mg + Fulvestrant | GS-5829 9 mg + Fulvestrant
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Randomized Phase 2 Dose Expansion: Clinical Benefit Rate
Description: Clinical benefit rate (CBR) was defined as the proportion of participants who achieve CR, PR, or stable disease that lasts for > 24 weeks based on RECIST v. 1.1 study progression criteria.
Time Frame: Baseline up to 2 years
Population: as for outcome 2
Arm/Group | GS-5829 4 mg + Exemestane | GS-5829 4 mg + Fulvestrant | GS-5829 6 mg + Fulvestrant | GS-5829 9 mg + Fulvestrant
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Randomized Phase 2 Dose Expansion: Overall Survival
Description: Overall survival was defined as the interval from date of randomization to date of death from any cause.
Time Frame: Baseline up to 2 years
Population: as for outcome 2
Arm/Group | GS-5829 4 mg + Exemestane | GS-5829 4 mg + Fulvestrant | GS-5829 6 mg + Fulvestrant | GS-5829 9 mg + Fulvestrant
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose date to last dose date (average: 14.5 weeks; maximum: 53 weeks) plus 30 days
Description: Safety Analysis Set included all participants who were enrolled and received at least 1 dose of any study drug.
Arm/Group | GS-5829 4 mg + Exemestane | GS-5829 4 mg + Fulvestrant | GS-5829 6 mg + Fulvestrant | GS-5829 9 mg + Fulvestrant
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 2/3 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GS-5829 4 mg + Exemestane (N=4) | GS-5829 4 mg + Fulvestrant (N=3) | GS-5829 6 mg + Fulvestrant (N=3) | GS-5829 9 mg + Fulvestrant (N=3)
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GS-5829 4 mg + Exemestane (N=4) | GS-5829 4 mg + Fulvestrant (N=3) | GS-5829 6 mg + Fulvestrant (N=3) | GS-5829 9 mg + Fulvestrant (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 1 | 3
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 2 | 1 | 1
Gait disturbance (General disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Injection site bruising (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Oral infection (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Breast haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol: Original (2016-06-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT02983604/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-08-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT02983604/Prot_001.pdf
  • Study Protocol: Amendment 2 (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT02983604/Prot_002.pdf
  • Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT02983604/SAP_003.pdf